Standing Committee for Research Ethics on Living Creatures Membership NO: HAP – 05 – D – 003, NCBE, KSA. Registration NO: IORG0006803, Office for Human Research Protections (OHRP), USA.





## INFORMED CONSENT STATEMENT

For children/minors participating in this study, the term "You" addresses both the participant and the parents or legally authorized representative to consent.

# PROJECT TITLE: The Efficacy of Non-invasive Brain Stimulation on Cognitive Functions in Patients with Chronic Obstructive Pulmonary Disease: Double-Blinded Randomised Controlled Trial

- Name of the Investigator/s-
  - Shahad Alkandari
  - Dr. Turki Abualait
  - Dr. Mohammad Al-Subaiei

## (Affiliation):

Imam Abdulrahman Bin Faisal University.

 You are being asked to participate in our study of Title the Association Between Cognitive Impairment and Chronic Obstruction Pulmonary Disease.

For the period/duration of 24 months.

You were particularly selected to participate in this study because you are eligible based on the inclusion criteria.

We are investigating this topic to further our understanding of the objectives of our work to investigate the efficacy of a novel intervention, which is noninvasive brain stimulation (NIBS), to improve the cognitive function in patients with COPD.

Your participation in the research study is voluntary. Before agreeing to be a part of this study please read and/or listen to the following information carefully.

# بيان الموافقة المسبقة المتبصرة

للأطفال والقاصرين المشاركين في هذه الدراسة، فإن مصطلح "أنت" يخاطب كل من المشاركين والوالدين أو من ينوب عنه قانونياً.

عنوان المشروع: فعالية تحفيز الدماغ غير الجراحي على الوظائف الإدراكية لدى مرضى الانسداد الرئوي المزمن: تجربة عشوائية محكومة مزدوجة التعمية

# أسماء الباحثين:

- شهد الكندرى
- دكتور تركى أبو عليط
- دكتور محمد السبيعي

(الجهة الأكاديمية):

جامعة الإمام عبدالرحمن بن فيصل

1. نحن نطلب منك أن تشارك في دراستنا

بعنوان: العلاقة بين الضعف الإدراكي ومرض الانسداد الرئوي المزمن

المدة /الفترة: 24 شهراً

تم اختيارك شخصياً لتشارك في هذه الدراسة لأن حالتك الصحية تتوافق مع متطلبات البحث

ونحن نبحث في هذا الموضوع من أجل زيادة فهمنا عن تقييم فعالية تدخل جديد، وهو تحفيز الدماغ غير الجراحي NIBS، لتحسين الوظيفة الإدراكية لدى مرضى الانسداد الرئوي المزمن.

يرجى ملاحظة أن مشاركتك في هذه الدراسة البحثية تعتبر تطوعية وقبل الموافقة على أن تكون جزءا من هذه الدراسة يرجى قراءة و / أو الاستماع

Standing Committee for Research Ethics on Living Creatures Membership NO: HAP – 05 – D – 003, NCBE, KSA. Registration NO: IORG0006803, Office for Human Research Protections (OHRP), USA.





Feel free to ask questions if you have any ambiguities.

- 2. If you participate in this study, you may be asked to donate a sample of blood which will be sent to the laboratory in King Fahad University Hospital for analysis. Your sample will be coded; however, investigators at the laboratory in King Fahad University Hospital will not have any access to your personal information and clinical data. You will also be required to answer some questions, which will be analyzed. Your answers will be coded, and researchers at Imam Abdulrahman bin Faisal University will not have access to your personal information and data. You will also be required to undergo medical tests such as ultrasound and physical fitness test under the supervision of qualified specialists. The test results will be analyzed, and the data will be confidential.
- In addition, the investigator will acquire clinical data from your medical record at the hospital.
- 4. Risks are limited to the usual discomfort of donating specific samples or discomfort of using NIBS as previous studies have proven that it is a safe device with no significant risks, and mild fatigue may be felt after the fitness tests.
- 5. This study designed might benefit you and other similar patients, besides", however, there is a possibility that the results of the study may contribute to future alternative treatments and procedures of [NIBS] that might also be beneficial.
- 6. All information obtained you're your medical records during the study will be confidential. Your privacy will be always protected. You will not be identified individually in any way

إلى المعلومات التالية بعناية ، لا تتردد في طرح الأسئلة إذا كان هناك شيء لم تفهمه.

- 2. إذا قمت بالشاركة في هذه الدراسة فقد يطلب منك التبرع بعينة دم والتي سيتم إرسالها مختبر مستشفى الملك فهد الجامعي لتحليلها. عينتك ستكون مشفرة والباحثين في مختبر مستشفى الملك فهد الجامعي لا يستطيعون الوصول إلى معلوماتك الشخصية وبياناتك السريرية. كما سيتطلب منك الإجابة على بعض الأسئلة والتي سيتم تحليلها. إجاباتك ستكون مشفرة والباحثين في جامعة الإمام عبدالرحمن بن فيصل لا يستطيعون الوصول إلى معلوماتك وبياناتك الشخصية.
  - كما سيتطلب منك عمل فحوصات طبية كالسونار وفحوصات لياقة بدنية تحت اشراف مختصين متمكنين. وسيتم تحليل نتائج الفحوصات وستكون البيانات سرية.
- بالإضافة إلى ذلك فإن الباحث سيحصل على البيانات السريرية من سجلك الطبي في المستشفى.
- 4. تقتصر المخاطر على عدم الراحة المعتادة من التبرع بعينة الدم أو عدم الراحة من استخدام جهاز NIBS حيث أثبتت الدراسات بأنه جهاز آمن بدون أخطار جسيمة تذكر ويمكن الإحساس بالتعب البسيط بعد فحوصات اللياقة البدنية.
- 5. تم تصميم هذه الدراسة لاحتمالية الفائدة لك وللمرضى المشابهين لحالتك. وكما أن نتائج الدراسة يحتمل استخدامها مستقبلاً في علاجات بطرق بديلة مثل NIBS التي يمكن أن تكون ذات فائدة.
- 6. إن جميع المعلومات التي تم الحصول عليها من السجلات الخاصة بك أثناء الدراسة سرية وستتم حماية خصوصيتك في جميع الأوقات ولن يتم التعرف عليك شخصيًا بأي شكل من الأشكال كنتيجة لشاركتك في هذه الدراسة. ومع ذلك فإن البيانات التي تم جمعها

Standing Committee for Research Ethics on Living Creatures Membership NO: HAP – 05 – D – 003, NCBE, KSA. Registration NO: IORG0006803, Office for Human Research Protections (OHRP), USA.





because of your participation in this research. The data collected, however, may be used as part of publications and papers related to [the research itself].

- 7. In case of any unexpected injury or harm during this study, compensation will be given as per the rules and regulations of the Imam Abdulrahman Bin Faisal university.
- 8. Your participation in this study is entirely voluntary. You have rights to discontinue or refuse to participate even after initiation of study at any time for any reason. Such a refusal will not have any negative consequences for you.
- 9. You can stop participating at any time for any reason and without any consequences.
- Feel free to ask any question about anything that seems unclear to you. Also, you should carefully consider this study and consent form before signing
- 11. After your participation, in case you have any questions and/or concerns about research, want clarification or report any matter related to your participation in the research you may contact (Shahad Alkandari) any time on the number (0591440882)or via email (2240700005@iau.edu.sa) In addition, if any new information is learnt, at any time during the research, which might affect your participation in the study, you shall be informed.
- 12. Principal Investigator of the study will also sign the copy of Informed consent, and the signed copy of the Informed Consent will be handed over to the Study Participant. Also, signed copy of informed consent must be kept in the PI file, SCRELC file, and patient's medical record file.

- 7. في حالة حدوث أي أذى أو ضرر غير متوقعة خلال هذه الدراسة سيتم تعويض ذلك من قبل جامعة الإمام عبدالرحمن بن فيصل حسب النظم واللوائح.
- 8. مشاركتك في هذه الدراسة تطوعية تمامًا ولك أن ترفض المشاركة في هذا البحث وهذا الرفض ليس له أي عواقب سلبية بالنسبة لك إذا كنت بدأت المشاركة في البحث.
- يمكنك التوقف عن المشاركة في أي وقت ولأي سبب من الأسباب
  ومن دون أى عواقب.
- 10. خذ الحرية ولا تتردد في طرح أي سؤال عن أي شيء يبدو غير واضح لك ولك أن تنظر بعناية لهذه الدراسة البحث ونموذج الموافقة قبل التوقيع.
- 11. بعد مشاركتك، وفي حالة لديك أي استفسار على البحث أو طلب إيضاح لأي موضوع فيمكنك التواصل مع السيدة (شهد الكندري) في أي وقت على الجوال رقم (224070005) أو البريد الإلكتروني ( 224070005@iau.edu.sa) هذا بالإضافة إلى أنه سيتم إبلاغك بأية معلومات تؤثر على مشاركتك أثناء تنفيذ البحث
- 12. يوقع الباحث الرئيس على نموذج الموافقة بعد التبصير، ونسخة من النموذج الموقع تعطى للمشارك. نسخة موقعة من الموافقة قبل التبصير يجب الاحتفاظ بها في ملف الباحث الرئيس وملف اللجنة الدائمة لأخلاقيات البحث على المخلوقات الحيَّة وملف السجل الطبى للمريض.

Standing Committee for Research Ethics on Living Creatures Membership NO: HAP – 05 – D – 003, NCBE, KSA. Registration NO: IORG0006803, Office for Human Research Protections (OHRP), USA.





I have read or listened to the above information, and I have decided that I will participate in the project as described above. The researcher has explained to me about the study, other beneficial treatments or procedures available and clarified my doubts. I also understand what will be expected of me. I now understand that the purpose of the study is to [investigate the efficacy of a novel intervention, which is noninvasive brain stimulation (NIBS), to improve the cognitive function in patients with COPD.]. If I do not participate, there will be no penalty or loss of rights. I can stop participating at any time, even after I have started.

لقد قرأت أو استمعت إلى المعلومات المذكورة أعلاه وعليه فقد قررت أنني سوف أشارك في المشروع المذكور. وأوضح الباحث الدراسة بالنسبة لي وأجاب على أسئلتي. وأنا واع تمامًا بما سيطلب مني. وأنا على يقين أن الغرض من هذه الدراسة هو [تقييم فعالية تدخل جديد، وهو تحفيز الدماغ غير الجراحي NIBS، لتحسين الوظيفة الإدراكية لدى مرضى الانسداد الرئوى المزمن.]

وإذا لم أشارك فلن تكون هناك عقوبة أو فقدان للحقوق ويمكنني التوقف عن المشاركة في أي وقت حتى بعد أن أكون قد بدأت فعليًا بالمشاركة.

I agree to participate in the study and for my samples to be kept and used for future research.

My signature below also indicates that I have received a copy of this English consent form together with an official translation of this document in Arabic.

Participant's signature

Principal Investigator signature

أوافق على المشاركة في هذه الدراسة ولا مانع من أن تحفظ عيناتي وتستخدم للبحث في المستقبل.

يشير توقيعي أدناه أيضا بأنني تلقيت نسخة من نموذج الموافقة باللغة العربية إلى جانب ترجمة رسمية لهذه الوثيقة باللغة الانجليزية.

توقيع المشارك:

وقيع الباحث الرئيسي: